CLINICAL TRIAL: NCT00565253
Title: Inhaled Nitric Oxide in Pulmonary Embolism, a Randomized, Double-Blind Placebo-Controlled Study
Brief Title: Inhaled Nitric Oxide in Pulmonary Embolism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 3052001
Record Dates: First submitted 2007-11-28; First posted 2007-11-29 (Estimated); Last update posted 2010-06-23 (Estimated); Status verified 2010-06

CONDITIONS: Pulmonary Embolism
Keywords: pulmonary embolism; inhaled nitric oxide
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Inhaled nitric oxide (NO) — 20 ppm for 15 minutes

SUMMARY:
The purpose of the study is to determine if inhaled nitric oxide, a potent and selective pulmonary vasodilator, is beneficial in patients with acute pulmonary embolism causing increased right ventricular afterload.

DETAILED DESCRIPTION:
The early phase of severe pulmonary embolism is associated with high mortality. Right ventricular failure induced by the increase in right ventricular afterload is the final cause of deterioration leading to circulatory failure in patients who die from severe pulmonary embolism. Therefore, reduction of right ventricular afterload remains the central therapeutic strategy. In acute pulmonary embolism, the increase in pulmonary vascular resistance is caused by reduction in the cross-sectional area of the pulmonary vascular bed from obstructing emboli. Pulmonary arterial constriction further increases pulmonary vascular resistance, whereby vasoactive humoral factors may be contributing, which are released from activated platelets accumulating at the site of the clot. Consequently, administration of vasodilators of the pulmonary circulation may be regarded as a therapeutic option to antagonize increased pulmonary vasoconstriction or compensate for impaired vasodilation. Inhaled nitric oxide (NO) acts as a powerful selective pulmonary vasodilator. The aim of the study is to determine, if short-term inhalation of NO is beneficial in respiratory compromised patients with right ventricular dysfunction after acute pulmonary embolism.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute pulmonary embolism within 24 hours after onset of symptoms.
* Patients with hypoxaemia not present before pulmonary embolism and acute right ventricular dysfunction.

Exclusion Criteria:

* Age < 18 years.
* Chronic lung disease, left heart failure, suspected or documented intracranial bleeding.
* Pregnancy, Methaemoglobinaemia.
* Patients who previously needed thrombolysis or surgical embolectomy.
* Negative D-Dimer test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-03; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
right ventricular size and arterial oxygenation | 2 hours

SECONDARY OUTCOMES:
blood pressure, central venous pressure, right ventricular function, pulmonary artery pressure | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schenk, Prof MD MSc, Principal Investigator — Dpt. of Internal Medicine III, Medical University Vienna, Austria
Locations (1):
- University of Emergency Medicine, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Background] Capellier G, Jacques T, Balvay P, Blasco G, Belle E, Barale F. Inhaled nitric oxide in patients with pulmonary embolism. Intensive Care Med. 1997 Oct;23(10):1089-92. doi: 10.1007/s001340050461. PMID 9407246
- See also: Related Info — http://www.ards.org/learnaboutards/treatment/nitricoxide.html